CLINICAL TRIAL: NCT02703922
Title: Evaluation of a Diagnostic Strategy for Giant Cell Arteritis Based on Color Doppler Ultrasound of Temporal Arteries
Brief Title: Validation of a Diagnostic Algorithm of Giant Cell Arteritis
Acronym: ECHORTON
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Collaborators: Groupe Hospitalier de la Rochelle Ré Aunis (Other); Centre Hospitalier de Rochefort (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ECHORTON
Record Dates: First submitted 2016-03-03; First posted 2016-03-09 (Estimated); Results first posted 2024-12-13 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-11

CONDITIONS: Giant Cell Arteritis
MeSH Terms: conditions — Giant Cell Arteritis | interventions — Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GCA suspicion (Other): A first screening is performed using color Doppler ultrasound. In case of negative results, patients undergo TAB.
  Interventions: Other: color Doppler ultrasound and TAB in case of CDU negative

INTERVENTIONS:
Other: color Doppler ultrasound and TAB in case of CDU negative — Screening with color Doppler ultrasound followed by TAB in case of CDU negative

SUMMARY:
Giant cell arteritis (GCA or temporal arteritis or cranial arteritis) or Horton disease is a vasculitis that occurs in older adults, affecting vessels of medium and large caliber. The diagnosis of GCA is a challenge for general practitioners and specialists. Since 1970, it is based on a combination of clinical, biological and histological signs. Temporal artery biopsy (TAB) was the reference method until recently. However, TAB has many drawbacks. Therefore, researches of the past 20 years have been intended to develop alternative diagnostic methods. This was notably the case of the color Doppler ultrasound (CDU) since the description by Wolfgang Schmidt of the halo sign. Although European and British recommendations put CDU as second line method, many authors suggest the possibility to do without TAB in many cases. In addition, many practitioners believe that it is not "ethical" to use an invasive unprofitable procedure like TAB, and have already been using CDU in their routine practice. However, no diagnostic algorithm validating this approach in a prospective series has been published to date. Therefore, the present study aim at validating a diagnostic algorithm of giant cell arteritis using color Doppler imaging of temporal arteries and cervicocephalic axes as first screening method.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 50 years
* C reactive protein (CRP) above normal
* Suspected of GCA according to clinician expertise and / or aortitis arteritis or of one or more arteries from the aorta imaging (CT angiography, magnetic resonance angiography or positron emission tomography TDM18FDG)
* Benefiting from Social Security or receiving it via a third party
* have given their participation agreement by understanding and accepting the constraints of the study

Exclusion Criteria:

* Received corticosteroid dose ≥ 20 mg of prednisone equivalent for more than 7 days in the month before inclusion
* Underwent temporal artery biopsy before color Doppler ultrasound
* History of GCA
* Terminal palliative phase or suffering from a disease or comorbidities such as life is involved in less than a year
* Patient with severe cognitive impairment
* Patient that can not be followed by the investigator for the duration of the study
* Refusal to participate in the study
* With enhanced protection (namely those deprived of liberty by a court or administrative order, patient staying in a health or social institution, under legal protection, and patients in emergencies)
* Pregnant or breastfeeding women, women of childbearing age who do not have effective contraception
* Participating in another clinical trial.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2016-08-29 (Actual); Primary Completion 2020-02-10 (Actual); Study Completion 2022-02-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Roncato, MD, Study Director — Groupe Hospitalier de la Rochelle Ré Aunis; Guillaume Denis, MD, Study Director — Centre Hospitalier de Rochefort
Locations (6):
- France (6):
  - Centre Hospitalier d'Angoulême, Angoulême
  - Groupe Hospitalier de la Rochelle Ré Aunis, La Rochelle
  - Centre Hospitalier Universitaire de Nantes, Nantes
  - Centre Hospitalier de Niort, Niort
  - Centre Hospitalier Universitaire de Poitiers, Poitiers
  - Centre Hospitalier de Rochefort, Rochefort

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Weyand CM, Goronzy JJ. Giant-cell arteritis and polymyalgia rheumatica. N Engl J Med. 2014 Oct 23;371(17):1653. doi: 10.1056/NEJMc1409206. No abstract available. PMID 25337759
- [Background] Smith JH, Swanson JW. Giant cell arteritis. Headache. 2014 Sep;54(8):1273-89. doi: 10.1111/head.12425. Epub 2014 Jul 18. PMID 25041449
- [Background] Petri H, Nevitt A, Sarsour K, Napalkov P, Collinson N. Incidence of giant cell arteritis and characteristics of patients: data-driven analysis of comorbidities. Arthritis Care Res (Hoboken). 2015 Mar;67(3):390-5. doi: 10.1002/acr.22429. PMID 25132663
- [Background] Calvo-Romero JM. Giant cell arteritis. Postgrad Med J. 2003 Sep;79(935):511-5. doi: 10.1136/pmj.79.935.511. PMID 13679546
- [Background] Roblot P. [When should Horton's disease be suspected?]. Rev Prat. 1999 Mar 15;49(6):593-7. French. PMID 10218393
- [Background] Baslund B, Helleberg M, Faurschou M, Obel N. Mortality in patients with giant cell arteritis. Rheumatology (Oxford). 2015 Jan;54(1):139-43. doi: 10.1093/rheumatology/keu303. Epub 2014 Aug 13. PMID 25122725
- [Background] Nuenninghoff DM, Hunder GG, Christianson TJ, McClelland RL, Matteson EL. Mortality of large-artery complication (aortic aneurysm, aortic dissection, and/or large-artery stenosis) in patients with giant cell arteritis: a population-based study over 50 years. Arthritis Rheum. 2003 Dec;48(12):3532-7. doi: 10.1002/art.11480. PMID 14674005
- [Background] Kermani TA, Warrington KJ, Crowson CS, Ytterberg SR, Hunder GG, Gabriel SE, Matteson EL. Large-vessel involvement in giant cell arteritis: a population-based cohort study of the incidence-trends and prognosis. Ann Rheum Dis. 2013 Dec;72(12):1989-94. doi: 10.1136/annrheumdis-2012-202408. Epub 2012 Dec 19. PMID 23253927
- [Background] Hunder GG, Bloch DA, Michel BA, Stevens MB, Arend WP, Calabrese LH, Edworthy SM, Fauci AS, Leavitt RY, Lie JT, et al. The American College of Rheumatology 1990 criteria for the classification of giant cell arteritis. Arthritis Rheum. 1990 Aug;33(8):1122-8. doi: 10.1002/art.1780330810. PMID 2202311
- [Background] Hunder GG. The early history of giant cell arteritis and polymyalgia rheumatica: first descriptions to 1970. Mayo Clin Proc. 2006 Aug;81(8):1071-83. doi: 10.4065/81.8.1071. PMID 16901030
- [Derived] Roncato C, Allix-Beguec C, Bourgade R, Becker F, Goujon JM, Denis G, Espitia O. Temporal artery biopsy and temporal artery ultrasound inter-rater agreement for the diagnosis of giant cell arteritis: an ancillary analysis from the multicentre prospective ECHORTON study. Rheumatol Int. 2025 Oct 27;45(11):260. doi: 10.1007/s00296-025-06009-9. PMID 41144031
- [Derived] Denis G, Espitia O, Allix-Beguec C, Dieval C, Lorcerie F, Gombert B, Pouget-Abadie X, Toquet C, Agard C, Raimbeau A, Gautier G, Goujon JM, Durand G, Thollot-Karolewicz C, Lormeau C, Grados A, Grenot-Mercier A, El-Khoury R, Riche A, Hospital F, Visee S, Auriault ML, Landron C, Martin M, Roncato C. Diagnostic Strategy Using Color Doppler Ultrasound of Temporal Arteries in Patients With High Clinical Suspicion of Giant Cell Arteritis : A Prospective Cohort Study. Ann Intern Med. 2024 Jun;177(6):729-737. doi: 10.7326/M23-3417. Epub 2024 May 7. PMID 38710093

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: from end of August 2016 to February 2020 Type of location: five public hospitals
Groups:
- CDU Positive: A first screening is performed using color Doppler ultrasound (CDU).
  "CDU Positive" refers to patients with a bilateral clear halo sign (defined as homogenous, hypoechoic wall thickening, well-delineated toward the luminal side, visible both in longitudinal and transverse planes located on the superficial temporal arteries, trunk or branches) detected by color Doppler ultrasound
- CDU Negative: A first screening is performed using color Doppler ultrasound (CDU).
  "CDU negative" refers to patient with no sign or a unilateral halo sign on the temporal artery.
Period: Overall Study
Arm/Group | CDU Positive | CDU Negative
Started | 73 | 92
Completed | 58 | 74
Not Completed | 15 | 18
Not completed — Death | 5 | 8
Not completed — Lost to Follow-up | 10 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CDU Positive | CDU Negative | Total
Number analyzed (Participants) | 73 | 92 | 165
Age, Continuous [Mean (Standard Deviation); unit: years] | 79.6 (7.8) | 78 (9.6) | 78.7 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 60 | 102
  Male | 31 | 32 | 63
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  France | 73 | 92 | 165

OUTCOME MEASURES:

1. Primary Outcome: Number of CDU False-positive Patients
Description: patients with an alternative diagnosis within 2 years of follow-up among patients considered with giant cell arteritis (GCA) on a clinico-biological suspicion + Doppler "positive."
Time Frame: after 2 years of follow-up
Population: Patients followed up at two years
Measure: Count of Participants; unit: Participants
Arm/Group | CDU Positive | CDU Negative
Number analyzed (Participants) | 73 | 92
Participants
  Patients diagnosed with giant cell arteritis | 73 | 63
  Alternative diagnosis | 0 | 29

2. Secondary Outcome: Rate of "Temporal Artery Biopsy Positive" Among "Negative or Doubtful CDU "
Description: Number of temporal artery biopsy (TAB) positive patients among patients with negative or doubtful CDU
Time Frame: within 1 month (during diagnostic algorithm)
Measure: Count of Participants; unit: Participants
Arm/Group | CDU Negative
Number analyzed (Participants) | 92
Participants
  TAB negative | 28
  TAB positive | 57
  Uninterpretable | 7

3. Secondary Outcome: Number of Patients With a Persistent Halo at Second CDU Examination
Description: Describe S3/S4 Halo changes, and study correlation between persistence and poorer clinical response
Time Frame: after 2 years of follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | CDU Positive
Number analyzed (Participants) | 73
Participants
  Stable | 9
  Improvement | 30
  No more Halo | 25
  Not done | 9

4. Secondary Outcome: Number of Correctly Interpreted TAB
Description: Reproducibility of TAB interpretation
Time Frame: 1 month (after second blind reading of histological specimen and doppler imaging)
Population: According to the diagnostic algorithm, only ultrasound-negative patients underwent temporal artery biopsy within 7 days after the ultrasound
Measure: Count of Participants; unit: Participants
Arm/Group | CDU Negative
Number analyzed (Participants) | 92
Participants
  First analysis: Negative | 58
  First analysis: Positive | 28
  First analysis: inconclusive | 6
  First analysis: Not available | 0
  Blinded expert analysis: Negative | 55
  Blinded expert analysis: Positive | 18
  Blinded expert analysis: inconclusive | 4
  Blinded expert analysis: Not available | 15

5. Secondary Outcome: Number of Correctly Interpreted CDU
Description: Reproducibility of CDU interpretation
Time Frame: 1 month (after second blind reading of histological specimen and doppler imaging)
Measure: Count of Participants; unit: Participants
Arm/Group | CDU Positive | CDU Negative
Number analyzed (Participants) | 73 | 92
Participants
  First analysis: Positive | 73 | 0
  First analysis: negative | 0 | 92
  First analysis: Not available | 0 | 0
  Blinded expert analysis: Positive | 42 | 3
  Blinded expert analysis: negative | 16 | 75
  Blinded expert analysis: Not available | 15 | 14

ADVERSE EVENTS:
Time Frame: Two years after inclusion
Description: This study concern patients with high clinical suspicion of GCA defined by 2 mandatory criteria that were age >50 and biological inflammatory syndrome with C-Reactive Protein elevation, and at least one of the following factors: abnormal temporal arteries, scalp hyperesthesia, jaw claudication, vision loss, pain in the shoulder girdle or pelvic girdle, unusual headache, impaired general condition, fever, or imaging positive result and absence of obvious differential diagnosis.
Groups:
- CDU Positive: A first screening is performed using color Doppler ultrasound (CDU). "CDU Positive" refers to patients with a bilateral clear halo sign (defined as homogenous, hypoechoic wall thickening, well-delineated toward the luminal side, visible both in longitudinal and transverse planes located on the superficial temporal arteries, trunk or branches) detected by color Doppler ultrasound resonance angiography and/or positron emission tomography and absence of obvious differential diagnosis.
Arm/Group | CDU Positive | CDU Negative
All-Cause Mortality (participants affected / at risk) | 5/73 | 8/92
Serious Adverse Events (participants affected / at risk) | 12/73 | 18/92
Other Adverse Events (participants affected / at risk) | 51/73 | 50/92
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CDU Positive (N=73) | CDU Negative (N=92)
Acute prostatitis (Renal and urinary disorders) | 1 (1) | 1 (1)
Aneamia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Aneurysm of abdominal aorta (Cardiac disorders) | 1 (1) | 0 (0)
Aortic dissection rupture (Cardiac disorders) | 0 (0) | 1 (1)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Carotid artery stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral vasculitis (Vascular disorders) | 0 (0) | 1 (1)
Cognitive disorders (Nervous system disorders) | 1 (1) | 1 (1)
Covid-19 respiratory infection (Infections and infestations) | 0 (0) | 1 (1)
Dental abscess (Infections and infestations) | 1 (1) | 0 (0)
Dysfunction kidney (Renal and urinary disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Faint (Nervous system disorders) | 0 (0) | 1 (1)
Femoral neck fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Fracture due to osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Fracture of vertebral column without mention of spinal cord injury (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Generalised chest pains (General disorders) | 0 (0) | 1 (1)
Hemithyroidectomy (Endocrine disorders) | 0 (0) | 1 (1)
High grade atrioventricular block (Cardiac disorders) | 1 (1) | 0 (0)
Hyponatraemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Ischemic colitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Joint arthroplasty (Surgical and medical procedures) | 1 (1) | 0 (0)
Kidney failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Leukemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lumbar vertebral fracture L1 (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myelodysplasia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Osteoporosis steroid-induced (Product Issues) | 0 (0) | 2 (2)
Pachymeningitis (Nervous system disorders) | 0 (0) | 1 (1)
Palsy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pneumopathy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Spondylodiscitis (Infections and infestations) | 0 (0) | 1 (1)
Stroke (Nervous system disorders) | 1 (1) | 1 (1)
Tongue necrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urticaria recurrent (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Venous obstruction (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CDU Positive (N=73) | CDU Negative (N=92)
Abnormal weight gain (General disorders) | 2 (2) | 5 (5)
Abscesses of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Acute kidney failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Adenoma (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Amaurosis (Eye disorders) | 0 (0) | 1 (1)
Amyotrophy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Aneamia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Anorexia (General disorders) | 1 (1) | 0 (0)
Antral gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Anxiodepressive syndrome (Psychiatric disorders) | 1 (1) | 0 (0)
Aortitis (Cardiac disorders) | 0 (0) | 1 (1)
Arnold neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Arteritic anterior ischaemic optic neuropathy (Eye disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (1) | 3 (3)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
Back ache (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Bateman's purpura senilis (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Belly ache (General disorders) | 0 (0) | 1 (1)
Bleeding piles (Vascular disorders) | 1 (1) | 0 (0)
Blepharitis unspecified (Eye disorders) | 0 (0) | 1 (1)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Bronchopneumopathy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Calf swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Carcinoma (Immune system disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (1)
Cervical pain (General disorders) | 1 (1) | 1 (1)
Chest pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic myelomonocytic leukemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Claudication of jaw muscles (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cognitive disorders (Nervous system disorders) | 1 (1) | 0 (0)
Coxarthrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cramps (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0)
C-reactive protein increased (General disorders) | 1 (1) | 3 (3)
Cushingoid facies (Endocrine disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Diabetes mellitus (Endocrine disorders) | 3 (3) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dry eyes (Eye disorders) | 1 (1) | 0 (0)
Dysaesthesia (Nervous system disorders) | 1 (1) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Edema (Blood and lymphatic system disorders) | 3 (3) | 2 (2)
Epistaxis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Erythematous eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Fall (General disorders) | 3 (3) | 0 (0)
Fatigue (General disorders) | 1 (1) | 2 (2)
Finger dislocation (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Fixed pigmented erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Flexor tendon rupture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Flu (Infections and infestations) | 0 (0) | 1 (1)
Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Gastric infection (Infections and infestations) | 1 (1) | 0 (0)
Giant cell arteritis relapse (Vascular disorders) | 1 (1) | 0 (0)
Glaucoma unspecified (Eye disorders) | 0 (0) | 1 (1)
Hallucination (Nervous system disorders) | 0 (0) | 1 (1)
Headache (General disorders) | 3 (3) | 2 (2)
Heart failure (Cardiac disorders) | 1 (1) | 0 (0)
Hematoma (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Hot flushes facial (General disorders) | 1 (1) | 0 (0)
Hypertension (Cardiac disorders) | 2 (2) | 0 (0)
Idiopathic midline granuloma (Immune system disorders) | 0 (0) | 1 (1)
Inflammatory rheumatism (Vascular disorders) | 1 (1) | 0 (0)
Insomnia (General disorders) | 1 (1) | 6 (6)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Joint prothesis removal (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Junctional tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Knee osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lens luxation (Eye disorders) | 0 (0) | 1 (1)
Lumbar pain syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lump excision (Surgical and medical procedures) | 1 (1) | 0 (0)
Lung nodule (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Memory disturbance (Nervous system disorders) | 2 (2) | 1 (1)
Monocytosis (Infections and infestations) | 1 (1) | 0 (0)
Muscle pains (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Mycosis (Infections and infestations) | 0 (0) | 1 (1)
Myeloproliferative disorder (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Myopathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neovascular glaucoma (Eye disorders) | 1 (1) | 0 (0)
Oesophageal dysphagia (General disorders) | 0 (0) | 1 (1)
Olecranon bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Optic ischaemic neuropathy (Eye disorders) | 1 (1) | 0 (0)
Orthostatic hypotension (Cardiac disorders) | 1 (1) | 0 (0)
Osteoarthritis of neck (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Pain in ankle (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pancreatic lesion (Gastrointestinal disorders) | 0 (0) | 1 (1)
Paresthesia (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral lipodystrophy (Product Issues) | 0 (0) | 1 (1)
Peripheral neuropathy (Nervous system disorders) | 0 (0) | 2 (2)
Pneumopathy (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Polymyalgia rheumatica (Vascular disorders) | 2 (2) | 0 (0)
Ptosis (Eye disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rheumatism (Vascular disorders) | 0 (0) | 1 (1)
Rheumatoid vasculitis (Vascular disorders) | 0 (0) | 1 (1)
Rib fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rupture of muscle non-traumatic (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Shoulder and hand pain (General disorders) | 1 (1) | 0 (0)
Situational anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Sleep apnea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sleep disorder (General disorders) | 2 (2) | 1 (1)
Spontaneous ecchymoses (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Subacromial bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
cataract (Surgical and medical procedures) | 1 (1) | 0 (0)
Sweating (General disorders) | 1 (1) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 1 (1)
Telogen effluvium (Endocrine disorders) | 1 (1) | 0 (0)
Thyroid nodule (nontoxic) (Endocrine disorders) | 0 (0) | 1 (1)
Thyroiditis (Endocrine disorders) | 0 (0) | 1 (1)
Tingling sensation (Nervous system disorders) | 2 (2) | 1 (1)
Tremor (Nervous system disorders) | 2 (2) | 2 (2)
Urinary tract infection (Infections and infestations) | 3 (3) | 0 (0)
Uveitis (Eye disorders) | 1 (1) | 0 (0)
Venous thrombosis (Vascular disorders) | 1 (1) | 1 (1)
Vertigo (Nervous system disorders) | 0 (0) | 2 (2)
Visual acutity reduced (Eye disorders) | 3 (3) | 0 (0)
Vitreous detachment (Eye disorders) | 0 (0) | 1 (1)
Wound (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Wound dehiscence (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-04): https://cdn.clinicaltrials.gov/large-docs/22/NCT02703922/Prot_SAP_000.pdf